CLINICAL TRIAL: NCT00217906
Title: A+ Asthma Early Intervention in Asthma Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 299; R18HL063333 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Behavioral: A+ Asthma early intervention program

SUMMARY:
This project will evaluate the effectiveness of a Head Start-based early intervention for designed to improve asthma management skill and practices of parents, pre-school children and Head Start staff.

DETAILED DESCRIPTION:
BACKGROUND:

While increased asthma morbidity and mortality have been observed across all ethnicities, results from several studies have found that asthma morbidity has increased disproportionately in low-income African American children. Elementary school-based asthma education programs have shown promise in improving asthma management, and reducing asthma morbidity in this high-risk population, however, the fastest growing asthma risk is associated with children young than six. By elementary age many parents and children with asthma have well-established patterns of inappropriate asthma management that may be difficult to change. To date, no research has examined the impact of early intervention for asthma management in low-income, high-risk children.

DESIGN NARRATIVE:

Head Start sites will be randomized to either a minimal intervention control group or the A+ Asthma early intervention program designed to educate and assist Head Start teachers and family service coordinators to: optimize classroom management of asthma, educate, facilitate and reinforce appropriate parental medical and behavioral management of asthma, and instruct, model and reinforce early asthma knowledge and age-appropriate skills for preschool age children.

The primary outcome that the study was designed to evaluate Head Start absences/days enrolled, determined by review of Head Start attendance records.

The secondary outcomes specified in the protocol are health care utilization (emergency department visits, hospitalizations, primary care visits), asthma symptoms (restricted activity, symptom-free days, day and nighttime symptoms), asthma medications, parents' asthma-related quality of life, and parent, child and teacher asthma knowledge and management practices.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Children aged 3 and 4 years who have asthma that is currently active

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-10; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Rand — Johns Hopkins University

REFERENCES:
- [Background] Paasche-Orlow MK, Riekert KA, Bilderback A, Chanmugam A, Hill P, Rand CS, Brancati FL, Krishnan JA. Tailored education may reduce health literacy disparities in asthma self-management. Am J Respir Crit Care Med. 2005 Oct 15;172(8):980-6. doi: 10.1164/rccm.200409-1291OC. Epub 2005 Aug 4. PMID 16081544